CLINICAL TRIAL: NCT03834506
Title: A Phase 3, Randomized, Double-blind Study of Pembrolizumab (MK-3475) Plus Docetaxel Plus Prednisone Versus Placebo Plus Docetaxel Plus Prednisone in Participants With Chemotherapy-naïve Metastatic Castration-Resistant Prostate Cancer (mCRPC) Who Have Progressed on a Next Generation Hormonal Agent (NHA) (KEYNOTE-921)
Brief Title: Study of Pembrolizumab (MK-3475) Plus Docetaxel Versus Placebo Plus Docetaxel in Chemotherapy-naïve Metastatic Castration-resistant Prostate Cancer (mCRPC) (MK-3475-921/KEYNOTE-921)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3475-921; MK-3475-921 (Other: MSD); KEYNOTE-921 (Other: MSD); JAPAC-CTI (Registry Identifier: 194831); 2018-004116-22 (EudraCT Number)
Record Dates: First submitted 2019-02-06; First posted 2019-02-08 (Actual); Results first posted 2023-06-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Prostatic Neoplasms
Keywords: Programmed Cell Death 1 (PD 1, PD-1); Programmed Cell Death 1 Ligand 1 (PDL 1, PD-L1); Programmed Cell Death 1 Ligand 2 (PDL 2, PD-L2)
MeSH Terms: conditions — Prostatic Neoplasms; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — pembrolizumab; Docetaxel; Prednisone; Saline Solution; Dexamethasone; Calcium Dobesilate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab+Docetaxel (Experimental): Participants receive pembrolizumab 200 mg by intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W) for up to a maximum of 35 cycles (approximately 2 years) PLUS docetaxel 75 mg/m^2 by IV infusion on Day 1 of each 21-day cycle (Q3W) for a maximum of 10 cycles (approximately 7 months). Participants also concomitantly receive dexamethasone 8 mg by oral tablets at 12 hours, 3 hours, and 1 hour prior to docetaxel administration and prednisone 5 mg by oral tablets twice daily during each 21-day docetaxel cycle.
  Interventions: Biological: Pembrolizumab; Drug: Docetaxel; Drug: Prednisone; Drug: Dexamethasone
- Placebo+Docetaxel (Placebo Comparator): Participants receive placebo by IV infusion on Day 1 of each 21-day cycle (Q3W) for up to a maximum of 35 cycles (approximately 2 years) PLUS docetaxel 75 mg/m^2 by IV infusion on Day 1 of each 21-day cycle (Q3W) for a maximum of 10 cycles (approximately 7 months). Participants also concomitantly receive dexamethasone 8 mg by oral tablets at 12 hours, 3 hours, and 1 hour prior to docetaxel administration and prednisone 5 mg by oral tablets twice daily during each 21-day docetaxel cycle.
  Interventions: Drug: Docetaxel; Drug: Prednisone; Drug: Placebo; Drug: Dexamethasone

INTERVENTIONS:
Biological: Pembrolizumab — IV infusion
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab+Docetaxel
Drug: Docetaxel — IV infusion
  Other Names: TAXOTERE®
Drug: Prednisone — Oral tablets
Drug: Placebo — IV infusion
  Other Names: Normal saline or dextrose infusion
  Arms: Placebo+Docetaxel
Drug: Dexamethasone — Oral tablets
  Other Names: DECADRON®

SUMMARY:
The purpose of this study is to assess the efficacy and safety of the combination of pembrolizumab (MK-3475) and docetaxel in the treatment of men with metastatic castration-resistant prostate cancer (mCRPC) who have not received chemotherapy for mCRPC but have progressed on or are intolerant to Next Generation Hormonal Agent (NHA).

There are two primary study hypotheses.

Hypothesis 1: The combination of pembrolizumab plus docetaxel plus prednisone is superior to placebo plus docetaxel plus prednisone with respect to Overall Survival (OS).

Hypothesis 2: The combination of pembrolizumab plus docetaxel plus prednisone is superior to placebo plus docetaxel plus prednisone with respect to Radiographic Progression-free Survival (rPFS) per Prostate Cancer Working Group (PCWG)-modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as assessed by blinded independent central review.

DETAILED DESCRIPTION:
With Amendment 6 (effective date: 29-Sep-2022), all participants will be unblinded and placebo treatment will be stopping. Participants who are deemed to be deriving clinical benefit from treatment may continue at the discretion of the investigator.

The global study for MK-3475-921 enrolled 1030 participants. Of the 1030 total participants enrolled in the global study, 21 were also enrolled in the China extension study for MK-3475-921 (NCT04907227).

ELIGIBILITY:
The main inclusion and exclusion criteria include but are not limited to the following:

Inclusion Criteria:

* Has histologically- or cytologically-confirmed adenocarcinoma of the prostate without small cell histology
* Has prostate cancer progression while on androgen deprivation therapy (or post bilateral orchiectomy) within 6 months prior to screening
* Has current evidence of metastatic disease documented by either bone lesions on bone scan and/or soft tissue disease by computed tomography/magnetic resonance imaging (CT/MRI)
* Has received prior treatment with one (but not more than one) NHA (eg, abiraterone acetate, enzalutamide, apalutamide, or darolutamide) for metastatic hormone-sensitive prostate cancer (mHSPC) or castration-resistant prostate cancer (CRPC) and either a) progressed through treatment OR b) has become intolerant of the drug
* Has ongoing androgen deprivation with serum testosterone <50 ng/dL (<2.0 nM)
* Participants receiving bone resorptive therapy (including, but not limited to, bisphosphonate or denosumab) must have been on stable doses prior to randomization
* Participants must agree to the following during the study treatment period and for at least 120 days after the last dose of pembrolizumab or for at least 180 days after the last dose of docetaxel (whichever is longer): Refrain from donating sperm PLUS Use contraception unless confirmed to be azoospermic (vasectomized or secondary to medical cause)
* Participants must agree to use male condom when engaging in any activity that allows for passage of ejaculate to another person of any sex
* Has provided newly obtained core or excisional biopsy (obtained within 12 months of screening) from soft tissue not previously irradiated (samples from tumors progressing in a prior site of radiation are allowed). Participants with bone only or bone predominant disease may provide a bone biopsy sample
* Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 assessed within 7 days of randomization

Exclusion Criteria:

* Has a known additional malignancy that is progressing or has required active treatment in the last 3 years
* Has an active autoimmune disease that has required systemic treatment in past 2 years
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy
* Has undergone major surgery including local prostate intervention (excluding prostate biopsy) within 28 days prior to randomization and not recovered adequately from the toxicities and/or complications
* Has a gastrointestinal disorder affecting absorption or is unable to swallow tablets/capsules
* Has an active infection (including tuberculosis) requiring systemic therapy
* Has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis
* Has known active human immunodeficiency virus (HIV), hepatitis B virus (HBV) or hepatitis C virus (HCV) infection
* Has known active central nervous system (CNS) metastases and/or carcinomatous meningitis
* Has severe hypersensitivity (≥Grade 3) to pembrolizumab and/or any of its excipients
* Has symptomatic congestive heart failure (New York Heart Association Class III or IV heart disease)
* Has had a prior anti-cancer monoclonal antibody (mAb) prior to randomization or who has not recovered (i.e., Grade ≤1 or at baseline) from AEs due to mAbs
* Has used herbal products that may have hormonal anti-prostate cancer activity and/or are known to decrease PSA levels (e.g. saw palmetto) prior to randomization
* Has received prior treatment with radium or other therapeutic radiopharmaceuticals for prostate cancer
* Has received prior therapy with an anti-programmed cell death-1 (anti-PD-1), anti-programmed cell death-ligand 1 (anti-PD-L1), or anti PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., cytotoxic T-lymphocyte-associated protein 4 [CTLA-4], OX-40, CD137)
* Has received prior treatment with docetaxel or another chemotherapy agent for mCRPC
* Has hypersensitivity to docetaxel or polysorbate 80
* Is currently receiving either strong or moderate inhibitors of cytochrome P450 (CYP)3A4 that cannot be discontinued for the duration of the study
* Has received prior targeted small molecule therapy or abiraterone acetate, enzalutamide, apalutamide, or darolutamide within 4 weeks prior to the first dose of study treatment, or has not recovered (i.e., Grade ≤1 or at baseline) from AEs due to a previously administered agent
* Has received prior radiotherapy to within 2 weeks of start of study treatment. Participants must have recovered from all radiation-related toxicities, not require corticosteroids, and not have had radiation pneumonitis
* Has received a live vaccine within 30 days prior to randomization
* Has received treatment with 5α reductase inhibitors (eg, finasteride or dutasteride), estrogens, and/or cyproterone within 4 weeks prior to randomization
* Has received prior treatment with ketoconazole for prostate cancer
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks prior to the first dose of study treatment
* Has a "superscan" bone scan
* Is expecting to conceive or father children within the projected duration of the study, starting with the screening visit through 120 days after the last dose of study treatment
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1030 (Actual)
Dates: Start 2019-05-02 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2023-07-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (215):
- United States (28):
  - University of South Alabama, Mitchell Cancer Institute ( Site 0065), Mobile, Alabama
  - St. Joseph Heritage Healthcare ( Site 0069), Fullerton, California
  - University of Southern California Norris Comprehensive Cancer Center ( Site 0061), Los Angeles, California
  - USC Norris Oncology Hematology Newport Beach ( Site 0093), Newport Beach, California
  - University of California San Francisco ( Site 0023), San Francisco, California
  - University of Colorado Cancer Center ( Site 0022), Aurora, Colorado
  - Yale Cancer Center ( Site 0038), New Haven, Connecticut
  - Moffitt Cancer Center ( Site 0080), Tampa, Florida
  - Georgia Cancer Center at Augusta University ( Site 0026), Augusta, Georgia
  - Mount Sinai Hospital Medical Center ( Site 0042), Chicago, Illinois
  - Methodist Hospital- Merriillville ( Site 0008), Merrillville, Indiana
  - Karmanos Cancer Institute ( Site 0077), Detroit, Michigan
  - Henry Ford Health System ( Site 0039), Detroit, Michigan
  - Cancer & Hematology Centers of Western Michigan ( Site 0013), Grand Rapids, Michigan
  - Washington University School of Medicine ( Site 0057), St Louis, Missouri
  - St. Vincent Frontier Cancer Center ( Site 0016), Billings, Montana
  - Nebraska Cancer Specialists ( Site 0034), Omaha, Nebraska
  - Comprehensive Cancer Centers of Nevada ( Site 0092), Las Vegas, Nevada
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 0004), Hackensack, New Jersey
  - Associated Medical Professionals of NY ( Site 0060), Syracuse, New York
  - Duke Cancer Center ( Site 0010), Durham, North Carolina
  - W. G. Bill Hefner VA Medical Center ( Site 0029), Salisbury, North Carolina
  - University Hospitals Cleveland Medical Center ( Site 0036), Cleveland, Ohio
  - Oregon Health Sciences University ( Site 0031), Portland, Oregon
  - Carolina Urologic Research Center ( Site 0070), Myrtle Beach, South Carolina
  - Inova Schar Cancer Institute ( Site 0006), Fairfax, Virginia
  - Virginia Cancer Institute ( Site 0052), Richmond, Virginia
  - Blue Ridge Cancer Care ( Site 0086), Roanoke, Virginia
- Argentina (9):
  - Centro de Oncologia e Investigacion Buenos Aires COIBA ( Site 1013), Berazategui, Buenos Aires
  - Instituto de Investigaciones Clinicas ( Site 1000), Mar del Plata, Buenos Aires
  - Centro de Diagnostico Urologico ( Site 1008), Buenos Aires, Buenos Aires F.D.
  - Hospital Britanico de Buenos Aires ( Site 1006), Buenos Aires, Buenos Aires F.D.
  - Sanatorio Parque ( Site 1002), Rosario, Santa Fe Province
  - Instituto de Investigaciones Metabolicas [Buenos Aires, Argentina] ( Site 1011), Buenos Aires
  - Hospital Aleman ( Site 1004), Buenos Aires
  - Instituto Medico Alexander Fleming ( Site 1010), Buenos Aires
  - CEMAIC ( Site 1014), Córdoba
- Australia (7):
  - St George Hospital ( Site 0157), Kogarah, New South Wales
  - Macquarie University ( Site 0151), Macquarie University, New South Wales
  - Port Macquarie Base Hospital ( Site 0153), Port Macquarie, New South Wales
  - Calvary Mater Newcastle ( Site 0148), Waratah, New South Wales
  - Redcliffe Hospital ( Site 0161), Redcliffe, Queensland
  - John Flynn Hospital & Medical Centre ( Site 0164), Tugun, Queensland
  - Hollywood Private Hospital ( Site 0163), Nedlands, Western Australia
- Austria (4):
  - Medizinische Universitat Graz ( Site 0374), Graz, Styria
  - Ordensklinikum Linz GmbH Elisabethinen ( Site 0373), Linz, Upper Austria
  - SCRI-CCCIT GesmbH ( Site 0371), Salzburg
  - Medizinische Universitaet Wien ( Site 0375), Vienna
- Brazil (5):
  - Hospital de Caridade de Ijui ( Site 1038), Ijuí, Rio Grande do Sul
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da Pucrs ( Site 1021), Porto Alegre, Rio Grande do Sul
  - Centro de Novos Tratamentos Itajai - Clinica de Neoplasias Litoral ( Site 1035), Itajaí, Santa Catarina
  - Hospital de Base de Sao Jose de Rio Preto ( Site 1022), São José do Rio Preto, São Paulo
  - A.C. Camargo Cancer Center ( Site 1026), São Paulo
- Canada (9):
  - Nova Scotia Health Authority QEII-HSC ( Site 0114), Halifax, Nova Scotia
  - Hamilton Health Sciences-Juravinski Cancer Centre ( Site 0116), Hamilton, Ontario
  - Grand River Hospital ( Site 0120), Kitchener, Ontario
  - Lakeridge Health ( Site 0117), Oshawa, Ontario
  - Sunnybrook Research Institute ( Site 0108), Toronto, Ontario
  - Princess Margaret Cancer Centre ( Site 0107), Toronto, Ontario
  - CHU de Quebec-Universite Laval-Hotel Dieu de Quebec ( Site 0103), Québec, Quebec
  - CIUSSS du Bas Saint Laurent - Hopital Regional de Rimouski ( Site 0102), Rimouski, Quebec
  - CIUSSS de l Estrie - CHUS - Centre Hosp. Univ. Sherbrooke ( Site 0105), Sherbrooke, Quebec
- Chile (6):
  - Fundacion Arturo Lopez Perez ( Site 1049), Santiago, Region M. de Santiago
  - Pontificia Universidad Catolica de Chile ( Site 1047), Santiago, Region M. de Santiago
  - Bradford Hill Centro de Investigaciones Clinicas ( Site 1044), Santiago, Region M. de Santiago
  - Centro Investigación del Cáncer James Lind ( Site 1041), Temuco, Región de la Araucanía
  - Rey y Oreilly Limitada ( Site 1048), Temuco, Región de la Araucanía
  - Centro de Investigaciones Clinicas Vina del Mar ( Site 1042), Viña del Mar, Región de Valparaíso
- China (15):
  - Peking University First Hospital ( Site 1303), Beijing, Beijing Municipality
  - The Fifth Medical Center of PLA General Hospital ( Site 1307), Beijing, Beijing Municipality
  - Beijing Cancer Hospital ( Site 1305), Beijing, Beijing Municipality
  - The First Affiliated Hospital of Xiamen University ( Site 1319), Xiamen, Fujian
  - Sun Yat Sen Memorial Hospital ( Site 1323), Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangzhou Medical University ( Site 1330), Guangzhou, Guangdong
  - Harbin Medical University Cancer Hospital ( Site 1326), Harbin, Heilongjiang
  - Henan Cancer Hospital ( Site 1321), Zhengzhou, Henan
  - Hubei Cancer Hospital ( Site 1329), Wuhan, Hubei
  - Hunan Cancer Hospital ( Site 1320), Changsha, Hunan
  - Nanjing Drum Tower Hospital ( Site 1312), Nanjing, Jiangsu
  - Fudan University Shanghai Cancer Center ( Site 1300), Shanghai, Shanghai Municipality
  - Zhongshan Hospital Fudan University ( Site 1301), Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Zhejiang University School of Medicine ( Site 1309), Hangzhou, Zhejiang
  - Zhejiang Provincial People's Hospital ( Site 1310), Hangzhou, Zhejiang
- Colombia (10):
  - Hospital Pablo Tobon Uribe ( Site 1066), Medellín, Antioquia
  - Biomelab S A S ( Site 1067), Barranquilla, Atlántico
  - Clinica de la Costa Ltda. ( Site 1073), Barranquilla, Atlántico
  - Instituto Nacional de Cancerologia E.S.E ( Site 1061), Bogotá, Bogota D.C.
  - Clinica Colsanitas S.A. Sede Clinica Universitaria Colombia ( Site 1062), Bogotá, Bogota D.C.
  - Sociedad de Oncología Y Hematología del Cesar S.A.S. ( Site 1068), Valledupar, Cesar Department
  - Oncomedica S.A. ( Site 1057), Montería, Departamento de Córdoba
  - Oncologos del Occidente S.A. ( Site 1072), Pereira, Risaralda Department
  - Centro Medico Imbanaco de Cali S.A ( Site 1064), Cali, Valle del Cauca Department
  - Hemato Oncologos S.A. ( Site 1065), Cali, Valle del Cauca Department
- France (18):
  - C.H. de Saint Quentin ( Site 0481), Saint-Quentin, Aisne
  - Clinique Sainte Anne ( Site 0431), Strasbourg, Alsace
  - Centre Jean Perrin ( Site 0434), Clermont-Ferrand, Auvergne
  - Centre Leon Berard ( Site 0422), Lyon, Auvergne
  - Institut Paoli Calmettes. ( Site 0419), Marseille, Bouches-du-Rhone
  - CHU Jean Minjoz ( Site 0423), Besançon, Doubs
  - CHU de Brest -Site Hopital Morvan ( Site 0441), Brest, Finistere
  - Institut Bergonie ( Site 0421), Bordeaux, Gironde
  - Institut Claudius Regaud IUCT Oncopole ( Site 0418), Toulouse, Haute-Garonne
  - Hopital Foch ( Site 0428), Suresnes, Hauts-de-Seine
  - Institut De Cancerologie De L Ouest ( Site 0448), Saint-Herblain, Loire-Atlantique
  - Centre Hospitalier Regional du Orleans ( Site 0430), Orléans, Loiret
  - Centre D Oncologie de Gentilly ( Site 0432), Nancy, Meurthe-et-Moselle
  - C.H.U. Lyon Sud ( Site 0436), Pierre-Bénite, Rhone
  - CHU Amiens Picardie Site Sud Amiens ( Site 0438), Amiens, Somme
  - Institut Gustave Roussy ( Site 0416), Villejuif, Val-de-Marne
  - Institut Sainte Catherine ( Site 0447), Avignon, Vaucluse
  - Institut Mutualiste Montsouris ( Site 0446), Paris
- Germany (12):
  - Universitaetsklinikum Freiburg - Medizinische Klinik ( Site 0304), Freiburg im Breisgau, Baden-Wurttemberg
  - Universitaetsklinikum in Mannheim ( Site 0314), Mannheim, Baden-Wurttemberg
  - Studienpraxis Urologie ( Site 0309), Nürtingen, Baden-Wurttemberg
  - Universitaetsklinik fuer Urologie ( Site 0307), Tübingen, Baden-Wurttemberg
  - Klinikum Rechts der Isar ( Site 0300), Munich, Bavaria
  - Universitaetsklinik der Paracelsus Medizinischen Privatuniversitaet ( Site 0318), Nuremberg, Bavaria
  - Universitaetsklinikum Wuerzburg ( Site 0302), Würzburg, Bavaria
  - Universitaetsklinikum Goettingen ( Site 0345), Göttingen, Lower Saxony
  - Uniklinik RWTH Aachen ( Site 0308), Aachen, North Rhine-Westphalia
  - Universitaetsklinikum des Saarlandes ( Site 0348), Homburg, Saarland
  - Universitaetsklinikum Jena ( Site 0305), Jena, Thuringia
  - Charite Universitaetsmedizin Berlin ( Site 0301), Berlin
- Ireland (3):
  - Cork University Hospital ( Site 0727), Cork
  - Tallaght University Hospital ( Site 0730), Dublin
  - Mid Western Cancer Centre ( Site 0728), Limerick
- Israel (8):
  - Assaf Harofeh MC ( Site 0547), Beer Yaakov-Zerifin
  - Soroka Medical Center ( Site 0548), Beersheba
  - Rambam Medical Center ( Site 0543), Haifa
  - Hadassah Ein Kerem Medical Center ( Site 0546), Jerusalem
  - Meir Medical Center ( Site 0544), Kfar Saba
  - Rabin Medical Center ( Site 0545), Petah Tikva
  - Chaim Sheba Medical Center ( Site 0541), Ramat Gan
  - Sourasky Medical Center ( Site 0542), Tel Aviv
- Italy (7):
  - Istituto Clinico Humanitas Research Hospital ( Site 0452), Rozzano, Milano
  - Azienda Ospedaliera Cannizzaro ( Site 0458), Catania
  - A.O. Universitaria di Modena ( Site 0454), Modena
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale ( Site 0457), Napoli
  - Azienda Ospedaliera San Camillo Forlanini ( Site 0455), Roma
  - Azienda Ospedaliera Santa Maria Terni ( Site 0456), Terni
  - Presidio Ospedaliero Santa Chiara ( Site 0451), Trento
- Japan (20):
  - National Cancer Center Hospital East ( Site 0702), Kashiwa, Chiba
  - Toho University Sakura Medical Center ( Site 0703), Sakura, Chiba
  - National Hospital Organization Shikoku Cancer Center ( Site 0716), Matsuyama, Ehime
  - Kanazawa University Hospital ( Site 0701), Kanazawa, Ishikawa-ken
  - Kitasato University Hospital ( Site 0705), Sagamihara, Kanagawa
  - Yokohama City University Medical Center ( Site 0706), Yokohama, Kanagawa
  - Nara Medical University Hospital ( Site 0715), Kashihara, Nara
  - Kindai University Hospital ( Site 0714), Sayama, Osaka
  - Osaka University Hospital ( Site 0713), Suita, Osaka
  - Saitama Medical University International Medical Center ( Site 0708), Hidaka, Saitama
  - Dokkyo Medical University Saitama Medical Center ( Site 0707), Koshigaya, Saitama
  - Hamamatsu University Hospital ( Site 0720), Hamamatsu, Shizuoka
  - Yamaguchi University Hospital ( Site 0717), Ube, Yamaguchi
  - Chiba Cancer Center ( Site 0704), Chiba
  - Kyushu University Hospital ( Site 0718), Fukuoka
  - University of Miyazaki Hospital ( Site 0721), Miyazaki
  - Nagasaki University Hospital ( Site 0719), Nagasaki
  - Toranomon Hospital ( Site 0711), Tokyo
  - Nippon Medical School Hospital ( Site 0709), Tokyo
  - Keio University Hospital ( Site 0710), Tokyo
- Netherlands (11):
  - Ziekenhuis Gelderse Vallei ( Site 0485), Ede, Gelderland
  - Radboud University Medical Center ( Site 0470), Nijmegen, Gelderland
  - VieCuri Medisch Centrum ( Site 0487), Venlo, Limburg
  - Jeroen Bosch Ziekenhuis ( Site 1200), 's-Hertogenbosch, North Brabant
  - Catharina Ziekenhuis ( Site 0472), Eindhoven, North Brabant
  - Antoni van Leeuwenhoek Ziekenhuis ( Site 0480), Amsterdam, North Holland
  - Ziekenhuis Hilversum ( Site 0466), Hilversum, North Holland
  - Ziekenhuisgroep Twente ( Site 0469), Hengelo, Overijssel
  - Medisch Centrum Leeuwarden ( Site 0477), Leeuwarden, Provincie Friesland
  - Reinier de Graaf Groep ( Site 0484), Delft, South Holland
  - Hagaziekenhuis ( Site 1201), The Hague, South Holland
- Russia (14):
  - Chelyabinsk Regional Clinical Oncological Dispensary ( Site 0565), Chelyabinsk, Chelyabinsk Oblast
  - Krasnoyarsk Regional Clinical Oncological Dispensary ( Site 0585), Krasnoyarsk, Krasnoyarsk Krai
  - SBIH City clinical hospital named after D.D. Pletniov ( Site 0575), Moscow, Moscow
  - Russian Scientific Center of Radiology ( Site 0559), Moscow, Moscow
  - Central Clinical Hospital with Polyclinic ( Site 0562), Moscow, Moscow
  - National Medical Research Radiological Center ( Site 0556), Moscow, Moscow
  - Volga District Medical Center Federal Medical and Biological Agency ( Site 0572), Nizhny Novgorod, Nizhny Novgorod Oblast
  - Omsk Clinical Oncology Dispensary ( Site 0568), Omsk, Omsk Oblast
  - SBHI Samara Regional Clinical Oncology Dispensary ( Site 0576), Samara, Samara Oblast
  - Leningrad Regional Oncology Center ( Site 0588), Saint Petersburg, Sankt-Peterburg
  - Clinical Research Center of specialized types medical care-Oncology ( Site 0570), Saint Petersburg, Sankt-Peterburg
  - Russian Scientific Center of Radiology and Surgical Technologies ( Site 0567), Saint Petersburg, Sankt-Peterburg
  - SPb SBHI City Clinical Oncological Dispensary ( Site 0571), Saint Petersburg, Sankt-Peterburg
  - Tomsk National Research Medical Center of Russian Academy of Sciences ( Site 0579), Tomsk, Tomsk Oblast
- South Korea (5):
  - National Cancer Center ( Site 0174), Goyang-si, Kyonggi-do
  - Seoul National University Bundang Hospital ( Site 0175), Seongnam-si, Kyonggi-do
  - Seoul National University Hospital ( Site 0171), Seoul
  - Asan Medical Center ( Site 0176), Seoul
  - Samsung Medical Center ( Site 0172), Seoul
- Spain (11):
  - Instituto Catalan de Oncologia - ICO ( Site 0330), L'Hospitalet de Llobregat, Barcelona
  - Hospital Consorci Sanitari Parc Tauli ( Site 0335), Sabadell, Barcelona
  - Hospital Universitario Marques de Valdecilla ( Site 0336), Santander, Cantabria
  - Hospital Josep Trueta ( Site 0321), Girona, Gerona
  - Hospital del Mar ( Site 0333), Barcelona
  - Hospital Clinic ( Site 0323), Barcelona
  - Hospital Universitario Ramon y Cajal ( Site 0328), Madrid
  - Hospital Clinico San Carlos ( Site 0324), Madrid
  - Hospital Universitario HM Sanchinarro ( Site 0322), Madrid
  - Hospital Universitario Virgen de la Victoria ( Site 0337), Málaga
  - Hospital Virgen del Rocio ( Site 0329), Seville
- Taiwan (5):
  - National Cheng Kung University Hospital ( Site 0134), Tainen, Tainan
  - China Medical University Hospital ( Site 0132), Taichung
  - Taichung Veterans General Hospital ( Site 0133), Taichung
  - National Taiwan University Hospital ( Site 0131), Taipei
  - Taipei Veterans General Hospital ( Site 0135), Taipei
- United Kingdom (8):
  - University Hospitals Bristol NHS Foundation Trust ( Site 0530), Bristol, Bristol, City of
  - Cambridge University Hospitals NHS Trust ( Site 0540), Cambridge, Cambridgeshire
  - Torbay Hospital ( Site 0532), Torquay, Devon
  - Weston Park Hospital ( Site 0539), Sheffield, England
  - Royal Marsden Hospital ( Site 0526), Sutton, England
  - Mount Vernon Cancer Centre ( Site 0536), Northwood, Hertfordshire
  - Barts Cancer Institute ( Site 0483), London, London, City of
  - University of North Midlands NHS Foundation Trust ( Site 0527), Stoke-on-Trent, Staffordshire

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Petrylak DP, Ratta R, Matsubara N, Korbenfeld E, Gafanov R, Mourey L, Todenhofer T, Gurney H, Kramer G, Bergman AM, Zalewski P, De Santis M, Armstrong AJ, Gerritsen W, Pachynski R, Byun SS, Retz M, Levesque E, McDermott R, Bracarda S, Manneh R, Levartovsky M, Li XT, Schloss C, Poehlein CH, Fizazi K. Pembrolizumab Plus Docetaxel Versus Docetaxel for Previously Treated Metastatic Castration-Resistant Prostate Cancer: The Randomized, Double-Blind, Phase III KEYNOTE-921 Trial. J Clin Oncol. 2025 May 10;43(14):1638-1649. doi: 10.1200/JCO-24-01283. Epub 2025 Mar 5. PMID 40043230
- [Derived] Petrylak DP, Ratta R, Gafanov R, Facchini G, Piulats JM, Kramer G, Flaig TW, Chandana SR, Li B, Burgents J, Fizazi K. KEYNOTE-921: Phase III study of pembrolizumab plus docetaxel for metastatic castration-resistant prostate cancer. Future Oncol. 2021 Sep;17(25):3291-3299. doi: 10.2217/fon-2020-1133. Epub 2021 Jun 8. PMID 34098744
- See also: Merck Clinical Trials Information — http://merckclinicaltrials.com/
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26073&tenant=MT_MSD_9011

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Of the 1030 participants randomized in the MK-3475-921 global study, 21 participants were also included in the China extension study for MK-3475-921 (NCT04907227).
Groups:
- Pembrolizumab + Docetaxel: Participants received pembrolizumab 200 mg by intravenous (IV) infusion on Day 1 of each 21-day cycle (Q3W) for up to a maximum of 35 cycles (approximately 2 years) PLUS docetaxel 75 mg/m^2 by IV infusion on Day 1 of each 21-day cycle (Q3W) for a maximum of 10 cycles (approximately 7 months). Participants also concomitantly received dexamethasone 8 mg by oral tablets at 12 hours, 3 hours, and 1 hour prior to docetaxel administration and prednisone 5 mg by oral tablets twice daily during each 21-day docetaxel cycle.
- Placebo + Docetaxel: Participants received placebo by IV infusion on Day 1 of each 21-day cycle (Q3W) for up to a maximum of 35 cycles (approximately 2 years) PLUS docetaxel 75 mg/m^2 by IV infusion on Day 1 of each 21-day cycle (Q3W) for a maximum of 10 cycles (approximately 7 months). Participants also concomitantly received dexamethasone 8 mg by oral tablets at 12 hours, 3 hours, and 1 hour prior to docetaxel administration and prednisone 5 mg by oral tablets twice daily during each 21-day docetaxel cycle.
Period: Overall Study
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Started | 515 | 515
Treated | 514 | 514
Completed | 0 | 0
Not Completed | 515 | 515
Not completed — Death | 336 | 326
Not completed — Withdrawal by Parent/Guardian | 1 | 1
Not completed — Withdrawal by Subject | 10 | 8
Not completed — Sponsor decision | 165 | 178
Not completed — Physician Decision | 3 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: The baseline analysis population consisted of all randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel | Total
Number analyzed (Participants) | 515 | 515 | 1030
Age, Continuous [Mean (Standard Deviation); unit: Years] | 69.9 (7.9) | 70.4 (7.1) | 70.1 (7.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 515 | 515 | 1030
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 79 | 77 | 156
  Not Hispanic or Latino | 402 | 393 | 795
  Unknown or Not Reported | 34 | 45 | 79
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 6 | 8 | 14
  Asian | 78 | 76 | 154
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 13 | 13 | 26
  White | 401 | 399 | 800
  More than one race | 15 | 18 | 33
  Unknown or Not Reported | 1 | 1 | 2
Prior Treatment with a Next Generation Hormonal Agent (NHA): Abiraterone Acetate [Count of Participants; unit: Participants] — Participants were stratified according to prior treatment with abiraterone acetate. Participants were eligible for the study if they had received prior treatment with a NHA (abiraterone acetate) for metastatic hormone-sensitive prostate cancer (mHSPC) or metastatic castration-resistant prostate cancer (CRPC) and either progressed after treatment or became intolerant of the drug.
  Participants
    Yes | 278 | 277 | 555
    No | 237 | 238 | 475
Type of Metastases at Baseline [Count of Participants; unit: Participants] — Participants were stratified by the type of metastases present at baseline determined by blinded independent central review. If the metastases were only in the bone the participants were categorized as bone only. If the metastases were not in the bone, but in the liver, participants were categorized as liver. All other participants were categorized as other.
  Participants
    Bone only | 268 | 239 | 507
    Liver | 34 | 33 | 67
    Other | 213 | 243 | 456
Eastern Cooperative Oncology Group (ECOG) Performance Status (PS) [Count of Participants; unit: Participants] — Participants were classified by ECOG PS defined as:
  ECOG=0: Fully active, able to carry out all pre-disease performance with no restriction; ECOG=1: Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature; ECOG=2: Ambulatory and capable of all self-care but unable to carry out work activities, up and about >50% of waking hours; ECOG=3: Capable of only limited self-care, confined to bed or chair >50% of waking hours; ECOG=4: Completely disabled, cannot carry out self-care, totally confined to bed or chair; ECOG=5: Dead
  Participants
    ECOG = 0 | 298 | 286 | 584
    ECOG = 1 | 212 | 227 | 439
    ECOG = 2 | 0 | 0 | 0
    ECOG = 3 | 0 | 0 | 0
    ECOG = 4 | 1 | 0 | 1
    ECOG = 5 | 0 | 0 | 0
    Missing | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time from randomization to death due to any cause. The OS was calculated using the product-limit Kaplan-Meier (K-M) method for censored data. Participants without documented death at the time of the analysis were censored at the date of the last follow-up.
Time Frame: Up to 36.5 months
Population: All randomized participants in the intent to treat population who had data available for analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 515 | 515
Months | 19.6 [18.2 to 20.9] | 19.0 [17.9 to 20.9]
Statistical Analysis 1: Comparison: Pembrolizumab + Docetaxel vs Placebo + Docetaxel; Test type: Superiority; p = 0.1677, Log Rank — One-sided p-value based on log-rank test stratified by prior treatment with a NHA (abiraterone acetate) and type of metastases at baseline; Hazard Ratio (HR) = 0.92, 95% CI 2-sided [0.78 to 1.09] — HR based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by prior treatment with a NHA (abiraterone acetate) and type of metastases at baseline

2. Primary Outcome: Radiographic Progression-free Survival (rPFS) Per Prostate Cancer Working Group (PCWG)-Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: rPFS was defined as the time from randomization to occurrence of: radiological tumor progression using RECIST 1.1 as assessed by BICR; progression of bone lesions using PCWG criteria; or death due to any cause. Radiological progression as per RECIST 1.1 was ≥20% increase in sum of diameters of target lesions and progression of existing non-target lesions. Progression of bone lesions by PCWG criteria was the appearance of ≥2 new bone lesions on bone scan, that have been confirmed to not represent tumor flare, and was persistent for ≥6 weeks. The rPFS was calculated using the product-limit K-M method for censored data. Participants without a rPFS event were censored at the date of last disease assessment.
Time Frame: Up to approximately 28 months
Population: All randomized participants in the intent to treat population who had data available for analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 515 | 515
Months | 8.6 [8.3 to 10.2] | 8.3 [8.2 to 8.5]
Statistical Analysis 1: Comparison: Pembrolizumab + Docetaxel vs Placebo + Docetaxel; Test type: Superiority; p = 0.0335, Log Rank — One-sided p-value based on log-rank test stratified by prior treatment with NHA (abiraterone acetate) and type of metastases at baseline; Hazard Ratio (HR) = 0.85, 95% CI 2-sided [0.71 to 1.01] — HR based on Cox regression model with Efron's method of tie handling with treatment as a covariate stratified by prior treatment with NHA (abiraterone acetate) and type of metastases at baseline

3. Secondary Outcome: Time to Initiation of the First Subsequent Anti-cancer Therapy (TFST)
Description: TFST was defined as the time from randomization to initiation of the first subsequent anti-cancer therapy or death; whichever occurred first. The TFST was calculated using the product-limit K-M method for censored data. Any participant not known to have further subsequent therapy or death was censored at the last known time that no subsequent new anti-cancer therapy was received.
Time Frame: Up to approximately 28 months
Population: All randomized participants in the intent to treat population who had data available for analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 515 | 515
Months | 10.7 [10.4 to 11.1] | 10.4 [9.7 to 11.1]
Statistical Analysis 1: Comparison: Pembrolizumab + Docetaxel vs Placebo + Docetaxel; Test type: Superiority; p = 0.0331, Log Rank — [p-value comment as in outcome 2, analysis 1]; Hazard Ratio (HR) = 0.86, 95% CI 2-sided [0.74 to 1.01] — [estimate comment as in outcome 2, analysis 1]

4. Secondary Outcome: Prostate-specific Antigen (PSA) Response Rate
Description: The Prostate-specific Antigen (PSA) response rate was the percentage of participants who had PSA response defined as a reduction in the PSA level from baseline by ≥50%. The reduction in PSA level was confirmed by an additional PSA evaluation performed ≥3 weeks from the original response. The analysis was performed on participants who had baseline PSA measurements.
Time Frame: Up to 36.5 months
Population: All randomized participants in the intent to treat population, who had a PSA measurement at baseline, and had data available for analysis
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 474 | 486
Percentage of participants | 44.5 [40.0 to 49.1] | 45.7 [41.2 to 50.2]

5. Secondary Outcome: Objective Response Rate (ORR) Per Prostate Cancer Working Group (PCWG)-Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: ORR was defined as the percentage of participants with complete response (CR: disappearance of all target lesions per RECIST 1.1; and no evidence of disease (NED) on bone scan per PCWG) or partial response (PR: at least a 30% decrease in the sum of diameters of target lesions per RECIST 1.1; and non-progressive disease, non-evaluable [NE], or NED on bone scan or CR with non-progressive disease or NE bone scan per PCWG).
Time Frame: Up to 36.5 months
Population: All randomized participants in the intent to treat population, with measurable disease at baseline, and had data available for analysis
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 203 | 221
Percentage of participants | 33.5 [27.0 to 40.4] | 35.3 [29.0 to 42.0]
Statistical Analysis 1: Comparison: Pembrolizumab + Docetaxel vs Placebo + Docetaxel; Test type: Other; p = 0.6545, Miettinen & Nurminen method — Based on Miettinen & Nurminen method stratified by prior treatment with a NHA (abiraterone acetate) and type of metastases at baseline; Percent Difference = -1.8, 95% CI 2-sided [-10.7 to 7.1] — Based on Miettinen & Nurminen method stratified by prior treatment with a NHA (abiraterone acetate) and type of metastases at baseline

6. Secondary Outcome: Duration of Response (DOR) Per Prostate Cancer Working Group (PCWG)-Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: DOR was the time from first documented evidence of complete response (CR: disappearance of all target lesions per RECIST 1.1; and no evidence of disease [NED] on bone scan per PCWG) or partial response (PR: ≥30% decrease in the sum of diameters of target lesions per RECIST 1.1; and non-progressive disease, non-evaluable [NE], or NED on bone scan or CR with non-progressive disease or NE bone scan per PCWG) until progressive disease (PD) or death. PD per RECIST 1.1 was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of at least 5 mm. PD per PCWG was the appearance of ≥2 new bone lesions on bone scan, that have been confirmed to not represent tumor flare and were persistent for ≥6 weeks. The DOR was calculated using the product-limit K-M method for censored data. If a participant had not progressed, the participant was censored at the date of last disease assessment.
Time Frame: Up to 36.5 months
Population: All randomized participants in the intent to treat population, who demonstrated a CR or PR, and had data available for analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 68 | 78
Months | 6.3 [6.1 to 7.8] | 6.2 [6.2 to 6.4]

7. Secondary Outcome: Time to Pain Progression (TTPP) as Assessed by Brief Pain Inventory-Short Form (BPI-SF) Item 3 ("Worst Pain in 24 Hours") and Opiate Analgesic Use Assessed by the Analgesic Quantification Algorithm (AQA) Score
Description: TTPP was the time from randomization to pain progression (PP) based on BPI-SF Item 3 and AQA score. BPI-SF assesses pain intensity; for item 3, participant responses to "Please rate your pain at its worst in the last 24 hours" are scored from 0 (no pain) to 10 (worst pain). A higher score indicates greater pain. AQA captures the intensity of analgesic use in pain management, scored from 0 (no analgesic) to 7 (strong opioid use). A higher score indicates higher intensity of analgesic use.
  For participants asymptomatic at baseline, PP was ≥2-point change from baseline in BPI-SF item 3 score OR initiation of opioid use. For participants symptomatic at baseline, PP was ≥2-point change from baseline in the BPI-SF Item 3 score, a score of ≥4 and no decrease in average opioid use OR any increase in opioid use (e.g., 1 point change in AQA score). TTPP was assessed by product-limit K-M method. Participants with >2 consecutive unevaluable visits were censored at the last evaluable assessment.
Time Frame: Up to 36.5 months
Population: All participants in the patient-reported outcomes (PRO) full analysis set who received ≥1 dose of study treatment and who had ≥1 PRO assessment available
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 507 | 502
Months | 21.1 [13.7 to NA] — NA= Upper limit not reached at time of data cut off due to insufficient number of participants with an event. | NA [13.8 to NA] — NA= Median and upper limit not reached at time of data cut off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Docetaxel vs Placebo + Docetaxel; Test type: Other; p = 0.6178, Log Rank; One-sided p-value based on log-rank test stratified by prior treatment with NHA (abiraterone acetate) and type of metastases at baseline; Hazard Ratio (HR) = 1.05, 95% CI 2-sided [0.77 to 1.43] — [estimate comment as in outcome 2, analysis 1]

8. Secondary Outcome: Time to First Symptomatic Skeletal-related Event (SSRE)
Description: SSRE was the time from randomization to the first symptomatic skeletal-related event defined as:
  1. Use of external-beam radiation therapy (EBRT) to prevent or relieve skeletal symptoms
  2. Occurrence of new symptomatic pathologic bone fracture (vertebral or non-vertebral)
  3. Occurrence of spinal cord compression
  4. Tumor-related orthopedic surgical intervention, whichever occurs first.
  The SSRE was calculated using the product-limit K-M method for censored data. Participants without symptomatic skeletal-related events were censored at the last evaluable assessment.
Time Frame: Up to 36.5 months
Population: All randomized participants in the intent to treat population who had data available for analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 515 | 515
Months | NA [NA to NA] — NA=Median and lower and upper limits not reached at time of data cut off due to insufficient number of participants with an event. | NA [NA to NA] — NA=Median and lower and upper limits not reached at time of data cut off due to insufficient number of participants with an event.
Statistical Analysis 1: Comparison: Pembrolizumab + Docetaxel vs Placebo + Docetaxel; Test type: Other; p = 0.9788, Log Rank; [statistical method as in outcome 7, analysis 1]; Hazard Ratio (HR) = 1.54, 95% CI 2-sided [1.01 to 2.33] — [estimate comment as in outcome 2, analysis 1]

9. Secondary Outcome: Time to Prostate-specific Antigen (PSA) Progression
Description: The time to PSA progression was the time from randomization to PSA progression. The PSA progression date was defined as the date of:
  1. ≥25% increase and ≥2 ng/mL above the nadir, confirmed by a second value ≥3 weeks later if there was PSA decline from baseline; OR
  2. ≥25% increase and ≥2 ng/mL increase from baseline beyond 12 weeks if there was no PSA decline from baseline
  Time to PSA progression was calculated using the product-limit K-M method for censored data. Participants without PSA progression were censored at the last evaluable assessment.
Time Frame: Up to 36.5 months
Population: as for outcome 4
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 515 | 515
Months | 6.9 [6.2 to 7.6] | 7.0 [6.3 to 7.6]
Statistical Analysis 1: Comparison: Pembrolizumab + Docetaxel vs Placebo + Docetaxel; Test type: Other; p = 0.2970, Log Rank; [statistical method as in outcome 7, analysis 1]; Hazard Ratio (HR) = 0.96, 95% CI 2-sided [0.82 to 1.12] — [estimate comment as in outcome 2, analysis 1]

10. Secondary Outcome: Time to Radiographic Soft Tissue Progression Per Soft Tissue Rules of Prostate Cancer Working Group (PCWG)-Modified Response Evaluation Criteria in Solid Tumors Version 1.1 (RECIST 1.1) as Assessed by Blinded Independent Central Review (BICR)
Description: The time to radiographic soft tissue progression was defined as the time from randomization to radiographic soft tissue progression per soft tissue rules of PCWG-modified RECIST 1.1 as assessed by BICR. Progression was defined as ≥20% increase in the sum of diameters of target lesions. In addition to the relative increase of 20%, the sum must also have demonstrated an absolute increase of ≥5 mm. The appearance of one or more new lesions was also considered progression. Time to radiographic soft tissue progression was calculated using the product-limit K-M method for censored data. Participants without radiographic soft tissue progression were censored at the last evaluable assessment.
Time Frame: Up to 36.5 months
Population: All randomized participants in the intent to treat population who had data available for analysis
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 515 | 515
Months | 12.4 [10.7 to 14.9] | 11.2 [10.4 to 12.5]
Statistical Analysis 1: Comparison: Pembrolizumab + Docetaxel vs Placebo + Docetaxel; Test type: Other; p = 0.2876, Log Rank; [statistical method as in outcome 7, analysis 1]; Hazard Ratio (HR) = 0.95, 95% CI 2-sided [0.78 to 1.15] — [estimate comment as in outcome 2, analysis 1]

11. Secondary Outcome: Number of Participants Who Experienced an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who experienced an AE is presented.
Time Frame: Up to approximately 30 months
Population: All participants who received ≥1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 514 | 514
Participants | 508 | 505

12. Secondary Outcome: Number of Participants Who Discontinued Study Treatment Due To an Adverse Event (AE)
Description: An AE was any untoward medical occurrence in a clinical study participant, temporally associated with the use of study intervention, whether or not considered related to the study intervention. An AE could therefore have been any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a study intervention. The number of participants who discontinued study treatment due to an AE is presented.
Time Frame: Up to approximately 27 months
Population: All participants who received ≥1 dose of study treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
Number analyzed (Participants) | 514 | 514
Participants | 150 | 115

ADVERSE EVENTS:
Time Frame: Up to approximately 48 months
Description: All-cause mortality: All randomized participants; AEs: all participants who received ≥1 dose of study treatment. Per protocol, disease progression of cancer under study was not considered an AE unless considered related to study drug. Therefore, Medical Dictionary for Regulatory Activities (MedDRA) preferred terms "Neoplasm progression", "Malignant neoplasm progression" and "Disease progression" not related to study drug are excluded as AEs.
Arm/Group | Pembrolizumab + Docetaxel | Placebo + Docetaxel
All-Cause Mortality (participants affected / at risk) | 343/515 | 329/515
Serious Adverse Events (participants affected / at risk) | 212/514 | 197/514
Other Adverse Events (participants affected / at risk) | 496/514 | 488/514
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Docetaxel (N=514) | Placebo + Docetaxel (N=514)
Anaemia (Blood and lymphatic system disorders) | 5 (5) | 5 (5)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 28 (34) | 22 (23)
Immune thrombocytopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Necrotic lymphadenopathy (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Neutropenia (Blood and lymphatic system disorders) | 6 (10) | 7 (8)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Angina pectoris (Cardiac disorders) | 0 (0) | 1 (1)
Aortic valve stenosis (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 4 (4)
Cardiac arrest (Cardiac disorders) | 1 (1) | 2 (2)
Cardiac failure (Cardiac disorders) | 6 (6) | 0 (0)
Cardiac failure acute (Cardiac disorders) | 0 (0) | 2 (2)
Cardiac failure chronic (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac ventricular thrombosis (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve incompetence (Cardiac disorders) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 3 (3) | 1 (1)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 1 (1)
Pericarditis (Cardiac disorders) | 0 (0) | 1 (1)
Sinus tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Stress cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Subendocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0)
Supraventricular tachycardia (Cardiac disorders) | 1 (1) | 2 (2)
Ventricular fibrillation (Cardiac disorders) | 0 (0) | 1 (1)
Hypoacusis (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Vertigo (Ear and labyrinth disorders) | 0 (0) | 1 (2)
Hypophysitis (Endocrine disorders) | 0 (0) | 1 (1)
Hypothyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Blindness unilateral (Eye disorders) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1)
Diplopia (Eye disorders) | 1 (1) | 0 (0)
Retinal artery occlusion (Eye disorders) | 0 (0) | 1 (1)
Retinal tear (Eye disorders) | 1 (1) | 0 (0)
Anal fissure (Gastrointestinal disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 4 (4) | 0 (0)
Constipation (Gastrointestinal disorders) | 3 (4) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 13 (13) | 9 (10)
Diverticular perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenal ulcer haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Duodenitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 2 (2) | 0 (0)
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Immune-mediated enterocolitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Intestinal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intestinal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Large intestine perforation (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (2) | 2 (2)
Neutropenic colitis (Gastrointestinal disorders) | 1 (1) | 1 (1)
Oesophageal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Oesophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oroantral fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Proctitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal haemorrhage (Gastrointestinal disorders) | 0 (0) | 1 (2)
Stomatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 1 (1)
Chest discomfort (General disorders) | 0 (0) | 1 (1)
Chest pain (General disorders) | 1 (1) | 1 (1)
Complication associated with device (General disorders) | 1 (1) | 0 (0)
Death (General disorders) | 2 (2) | 2 (2)
General physical health deterioration (General disorders) | 2 (2) | 2 (2)
Inflammation (General disorders) | 1 (1) | 0 (0)
Mucosal inflammation (General disorders) | 1 (1) | 0 (0)
Multiple organ dysfunction syndrome (General disorders) | 1 (1) | 0 (0)
Oedema (General disorders) | 0 (0) | 1 (1)
Oedema peripheral (General disorders) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1)
Pyrexia (General disorders) | 6 (7) | 4 (4)
Autoimmune hepatitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hypertransaminasaemia (Hepatobiliary disorders) | 2 (2) | 0 (0)
Liver disorder (Hepatobiliary disorders) | 2 (2) | 0 (0)
Contrast media allergy (Immune system disorders) | 0 (0) | 1 (1)
Haemophagocytic lymphohistiocytosis (Immune system disorders) | 1 (1) | 0 (0)
Hypersensitivity (Immune system disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 1 (1) | 0 (0)
Abscess limb (Infections and infestations) | 1 (1) | 0 (0)
Abscess neck (Infections and infestations) | 1 (1) | 2 (2)
Anal abscess (Infections and infestations) | 2 (2) | 0 (0)
Appendicitis perforated (Infections and infestations) | 0 (0) | 1 (1)
Atypical pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Bacteraemia (Infections and infestations) | 1 (1) | 1 (1)
Bacterial infection (Infections and infestations) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 6 (6)
COVID-19 pneumonia (Infections and infestations) | 5 (5) | 6 (6)
Catheter site cellulitis (Infections and infestations) | 1 (1) | 0 (0)
Catheter site infection (Infections and infestations) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 2 (2) | 3 (3)
Clostridial sepsis (Infections and infestations) | 0 (0) | 1 (1)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 1 (1)
Cystitis (Infections and infestations) | 0 (0) | 1 (1)
Device related bacteraemia (Infections and infestations) | 0 (0) | 1 (1)
Device related infection (Infections and infestations) | 0 (0) | 1 (1)
Device related sepsis (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 0 (0) | 2 (2)
Encephalitis (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis (Infections and infestations) | 1 (1) | 0 (0)
Endophthalmitis (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 1 (1) | 0 (0)
Erysipelas (Infections and infestations) | 0 (0) | 1 (1)
Escherichia infection (Infections and infestations) | 1 (1) | 0 (0)
Gastroenteritis (Infections and infestations) | 0 (0) | 2 (2)
Gastroenteritis viral (Infections and infestations) | 1 (1) | 0 (0)
Herpes zoster meningomyelitis (Infections and infestations) | 1 (1) | 0 (0)
Infection (Infections and infestations) | 1 (1) | 2 (2)
Influenza (Infections and infestations) | 1 (1) | 0 (0)
Joint abscess (Infections and infestations) | 1 (1) | 0 (0)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 2 (2)
Meningitis meningococcal (Infections and infestations) | 0 (0) | 1 (1)
Meningoencephalitis herpetic (Infections and infestations) | 1 (1) | 0 (0)
Neutropenic sepsis (Infections and infestations) | 0 (0) | 1 (1)
Oropharyngeal candidiasis (Infections and infestations) | 0 (0) | 1 (1)
Parotitis (Infections and infestations) | 0 (0) | 1 (1)
Peritonitis (Infections and infestations) | 0 (0) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Pleural infection (Infections and infestations) | 1 (1) | 0 (0)
Pneumocystis jirovecii pneumonia (Infections and infestations) | 2 (2) | 0 (0)
Pneumonia (Infections and infestations) | 14 (14) | 12 (14)
Pneumonia bacterial (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia influenzal (Infections and infestations) | 0 (0) | 1 (1)
Pneumonia pneumococcal (Infections and infestations) | 0 (0) | 2 (2)
Pseudomembranous colitis (Infections and infestations) | 0 (0) | 2 (2)
Pyelonephritis (Infections and infestations) | 3 (3) | 2 (2)
Pyelonephritis acute (Infections and infestations) | 0 (0) | 3 (3)
Respiratory tract infection (Infections and infestations) | 1 (2) | 2 (2)
Rhinovirus infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 3 (3)
Septic shock (Infections and infestations) | 1 (1) | 2 (2)
Soft tissue infection (Infections and infestations) | 0 (0) | 1 (1)
Spinal cord infection (Infections and infestations) | 0 (0) | 1 (1)
Streptococcal infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 8 (8) | 7 (8)
Urinary tract infection bacterial (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Urosepsis (Infections and infestations) | 2 (2) | 4 (4)
Vascular device infection (Infections and infestations) | 1 (1) | 1 (1)
Vestibular neuronitis (Infections and infestations) | 1 (1) | 0 (0)
Acetabulum fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Cystitis radiation (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Femur fracture (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Fracture displacement (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Lower limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 (1) | 2 (2)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Pulmonary radiation injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Radiation proctitis (Injury, poisoning and procedural complications) | 1 (2) | 0 (0)
Rib fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Spinal fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (3)
Sternal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Transfusion related complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Alanine aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 0 (0)
Blood calcium increased (Investigations) | 0 (0) | 1 (1)
Blood creatinine increased (Investigations) | 1 (1) | 0 (0)
Hepatic enzyme increased (Investigations) | 1 (1) | 0 (0)
Influenza A virus test positive (Investigations) | 1 (1) | 0 (0)
Neutrophil count decreased (Investigations) | 4 (4) | 1 (1)
White blood cell count decreased (Investigations) | 1 (1) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Electrolyte imbalance (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 1 (1) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypervolaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypocalcaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hyponatraemia (Metabolism and nutrition disorders) | 3 (3) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Arthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 5 (6) | 6 (7)
Bone pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Crowned dens syndrome (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3)
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Myositis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (4)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Pathological fracture (Musculoskeletal and connective tissue disorders) | 6 (6) | 1 (1)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spinal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Adenocarcinoma gastric (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Adenocarcinoma of colon (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Bladder transitional cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Neuroendocrine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Small cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Tumour compression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Cauda equina syndrome (Nervous system disorders) | 0 (0) | 1 (1)
Cerebellar haematoma (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 3 (3) | 1 (1)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 1 (1) | 1 (1)
Lumbar radiculopathy (Nervous system disorders) | 1 (1) | 0 (0)
Myasthenia gravis (Nervous system disorders) | 1 (1) | 0 (0)
Nerve compression (Nervous system disorders) | 0 (0) | 1 (1)
Peripheral sensory neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Spinal cord compression (Nervous system disorders) | 1 (1) | 5 (5)
Subarachnoid haemorrhage (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 1 (1)
Device occlusion (Product Issues) | 1 (1) | 0 (0)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0)
Depression (Psychiatric disorders) | 1 (1) | 2 (2)
Acute kidney injury (Renal and urinary disorders) | 6 (6) | 3 (3)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1)
Calculus urinary (Renal and urinary disorders) | 1 (1) | 0 (0)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 1 (1)
Haematuria (Renal and urinary disorders) | 8 (9) | 4 (5)
Hydronephrosis (Renal and urinary disorders) | 0 (0) | 2 (2)
Renal failure (Renal and urinary disorders) | 1 (1) | 2 (2)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 1 (1) | 2 (2)
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Oedema genital (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (4)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Immune-mediated lung disease (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 5 (5) | 0 (0)
Lung disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Obstructive airways disorder (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 15 (15) | 6 (6)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 8 (8)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary toxicity (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 1 (1)
Stevens-Johnson syndrome (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arteriosclerosis (Vascular disorders) | 0 (0) | 1 (1)
Embolism (Vascular disorders) | 2 (2) | 2 (2)
Femoral artery aneurysm (Vascular disorders) | 0 (0) | 1 (2)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
Jugular vein thrombosis (Vascular disorders) | 0 (0) | 1 (1)
Orthostatic hypotension (Vascular disorders) | 2 (2) | 1 (1)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1)
Peripheral artery occlusion (Vascular disorders) | 0 (0) | 1 (1)
Venous thrombosis limb (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pembrolizumab + Docetaxel (N=514) | Placebo + Docetaxel (N=514)
Anaemia (Blood and lymphatic system disorders) | 147 (177) | 126 (168)
Neutropenia (Blood and lymphatic system disorders) | 41 (52) | 37 (47)
Hypothyroidism (Endocrine disorders) | 35 (37) | 16 (17)
Lacrimation increased (Eye disorders) | 33 (35) | 38 (38)
Abdominal pain (Gastrointestinal disorders) | 26 (30) | 28 (32)
Constipation (Gastrointestinal disorders) | 110 (152) | 85 (99)
Diarrhoea (Gastrointestinal disorders) | 209 (356) | 184 (289)
Nausea (Gastrointestinal disorders) | 124 (178) | 135 (194)
Stomatitis (Gastrointestinal disorders) | 34 (43) | 29 (30)
Vomiting (Gastrointestinal disorders) | 50 (70) | 70 (90)
Asthenia (General disorders) | 132 (180) | 128 (201)
Fatigue (General disorders) | 183 (255) | 184 (224)
Mucosal inflammation (General disorders) | 26 (31) | 31 (34)
Oedema peripheral (General disorders) | 95 (105) | 106 (120)
Pyrexia (General disorders) | 58 (69) | 42 (52)
Urinary tract infection (Infections and infestations) | 36 (48) | 33 (38)
Alanine aminotransferase increased (Investigations) | 27 (38) | 28 (30)
Aspartate aminotransferase increased (Investigations) | 29 (32) | 24 (27)
Blood alkaline phosphatase increased (Investigations) | 28 (28) | 25 (26)
Neutrophil count decreased (Investigations) | 47 (107) | 49 (112)
Weight decreased (Investigations) | 42 (45) | 29 (29)
White blood cell count decreased (Investigations) | 32 (60) | 27 (54)
Decreased appetite (Metabolism and nutrition disorders) | 107 (145) | 98 (126)
Hyperglycaemia (Metabolism and nutrition disorders) | 47 (54) | 54 (67)
Hypokalaemia (Metabolism and nutrition disorders) | 27 (37) | 15 (20)
Arthralgia (Musculoskeletal and connective tissue disorders) | 86 (125) | 99 (122)
Back pain (Musculoskeletal and connective tissue disorders) | 91 (105) | 101 (117)
Bone pain (Musculoskeletal and connective tissue disorders) | 44 (47) | 45 (51)
Myalgia (Musculoskeletal and connective tissue disorders) | 49 (55) | 42 (50)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 40 (47) | 46 (57)
Dizziness (Nervous system disorders) | 38 (42) | 41 (49)
Dysgeusia (Nervous system disorders) | 73 (88) | 79 (85)
Headache (Nervous system disorders) | 38 (49) | 34 (39)
Neuropathy peripheral (Nervous system disorders) | 27 (28) | 27 (30)
Peripheral sensory neuropathy (Nervous system disorders) | 132 (143) | 100 (108)
Insomnia (Psychiatric disorders) | 43 (51) | 46 (46)
Haematuria (Renal and urinary disorders) | 23 (25) | 28 (32)
Cough (Respiratory, thoracic and mediastinal disorders) | 47 (53) | 36 (39)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 61 (66) | 59 (63)
Alopecia (Skin and subcutaneous tissue disorders) | 182 (185) | 193 (198)
Dry skin (Skin and subcutaneous tissue disorders) | 23 (24) | 29 (32)
Nail discolouration (Skin and subcutaneous tissue disorders) | 25 (26) | 27 (28)
Nail disorder (Skin and subcutaneous tissue disorders) | 30 (30) | 30 (30)
Pruritus (Skin and subcutaneous tissue disorders) | 46 (53) | 26 (31)
Rash (Skin and subcutaneous tissue disorders) | 57 (70) | 54 (62)
Hypertension (Vascular disorders) | 28 (31) | 29 (32)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If publication activity is not directed by the Sponsor, the investigator agrees to submit all manuscripts or abstracts to the Sponsor before submission. This allows the Sponsor to protect proprietary information and to provide comments. Authorship will be determined by mutual agreement and in line with International Committee of Medical Journal Editors authorship requirements.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-09-29): https://cdn.clinicaltrials.gov/large-docs/06/NCT03834506/Prot_SAP_000.pdf